CLINICAL TRIAL: NCT00295061
Title: Multi-center, Randomized, Double-blind, Crossover Trial to Evaluate the Pharmacokinetic Comparability of Alpha-1 MP to Prolastin in Subjects With Alpha1-antitrypsin Deficiency.
Brief Title: Comparison of Pharmacokinetic, Safety, Tolerability of Alpha-1 MP and Prolastin In Alpha1-antitrypsin Deficient Adults
Acronym: ChAMP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Gerald Klein, MD, Chief Medical Officer, Vice President of Medical and Clinical Affairs, Talecris Biotherapeutics, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11816
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-08

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: alpha 1-Antitrypsin Deficiency; alpha 1-Antitrypsin; pulmonary emphysema
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Pulmonary Emphysema | interventions — Mp alpha1 receptor; alpha 1-Antitrypsin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Alpha-1 MP (Experimental): Sequential, blinded treatment periods of Alpha-1 MP (experimental), then crossed-over to Prolastin (active comparator), followed by open-label Alpha-1 MP
  Interventions: Drug: Alpha-1 MP
- 2 Prolastin (Active Comparator): Sequential, blinded treatment periods of Prolastin (active comparator), then crossed-over to Alpha-1 MP (experimental), followed by open-label Alpha-1 MP
  Interventions: Drug: alpha-1 proteinase inhibitor (human)

INTERVENTIONS:
Drug: Alpha-1 MP — alpha-1 proteinase inhibitor (human), 60 mg/kg body weight
  Other Names: Alpha-1 antitrypsin (AAT); TAL6004
  Arms: 1 Alpha-1 MP
Drug: alpha-1 proteinase inhibitor (human) — Prolastin
  Other Names: Alpha-1 antitrypsin (AAT); BAY x 5747; BAY 10-5233; TAL-05-00007
  Arms: 2 Prolastin

SUMMARY:
The purpose of this clinical study (ChAMP - Comparability pharmacokinetics of Alpha-1 Modified Process) is to compare the pharmacokinetic, safety and tolerability of Alpha-1 Proteinase Inhibitor (Human), modified process (Alpha-1 MP) and Prolastin in adult Alpha1-antitrypsin deficient patients. Patients will be infused intravenously with study drug on a weekly schedule for 24 weeks.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate the pharmacokinetic comparability of Alpha-1 MP to Prolastin® in subjects with Alpha1-antitrypsin deficiency.

This study is divided into three 8-week treatment sequences including an initial 8-week double-blind treatment period (with one of the 2 study drugs), a second 8-week double-blind treatment period (with the other study drug), and a third 8-week open-label treatment period (with Alpha-1 MP).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of congenital Alpha1-antitrypsin deficiency
* Must be receiving augmentation therapy with plasma-derived (human) Alpha1-Proteinase Inhibitor (Prolastin®) for at least one month prior to study entry.
* Signed written informed consent prior to initiation of any study related procedures

Exclusion Criteria:

* Females who are pregnant, breast feeding, or if of child-bearing potential, unwilling to practice adequate contraception throughout the study
* Use of systemic steroids within the 2 weeks prior to receiving study treatment (this does not include the use of inhaled steroids used on a routine or as needed basis).
* Subjects who have had exacerbations of their disease within one month of trial entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-05; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Hanna, MSc, Study Director — Grifols Therapeutics LLC
Locations (8):
- United States (8):
  - National Jewish Medical and Research Center, Denver, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - St Lukes-Roosevelt Hospital Center, New York, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Center at Tyler, Tyler, Texas

REFERENCES:
- [Derived] Stocks JM, Brantly ML, Wang-Smith L, Campos MA, Chapman KR, Kueppers F, Sandhaus RA, Strange C, Turino G. Pharmacokinetic comparability of Prolastin(R)-C to Prolastin(R) in alpha(1)-antitrypsin deficiency: a randomized study. BMC Clin Pharmacol. 2010 Sep 30;10:13. doi: 10.1186/1472-6904-10-13. PMID 20920295
- See also: The "Alpha-1 Foundation", dedicated to providing the leadership and resources that will result in increased research, improved health, worldwide detection and a cure for Alpha-1 Antitrypsin Deficiency — http://www.alphaone.org
- See also: AlphaNet, Inc devoted to improving the lives of individuals with Alpha-1 antitrypsin deficiency through comprehensive disease management services, clinical research administration, and consultative services — http://www.alphanet.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First-subject-first-dose was on 22 May 2006, Last-subject-last-visit was on 28 Feb 2007. The trial was performed at 6 clinical sites in the United States.
Groups:
- Alpha-1 MP / Prolastin: Sequential, blinded treatment periods of Alpha-1 modified process (MP) (experimental), then crossed-over to Prolastin (active comparator), followed by open-label Alpha-1 MP
- Prolastin / Alpha-1 MP: Sequential, blinded treatment periods of Prolastin (active comparator), then crossed-over to Alpha-1 MP (experimental), followed by open-label Alpha-1 MP
Period: Overall Study
Arm/Group | Alpha-1 MP / Prolastin | Prolastin / Alpha-1 MP
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Alpha-1 MP / Prolastin: Sequential, blinded treatment periods of Alpha-1 MP (experimental), then crossed-over to Prolastin (active comparator), followed by open-label Alpha-1 MP
- Total: Total of all reporting groups
Arm/Group | Alpha-1 MP / Prolastin | Prolastin / Alpha-1 MP | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (6.86) | 57.0 (9.33) | 57.7 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Alpha-1 MP vs. Prolastin® of Area Under the Curve (AUC) From Day 0 to Day 7
Description: The primary objective of this study was to demonstrate the pharmacokinetic comparability (geometric least square mean ratio of AUC between the Alpha-1 MP vs. Prolastin®, 90% confidence interval falls within 0.80-1.25, FDA Guidance as being "bioequivalent" between two treatments) of Alpha-1 MP to Prolastin® in subjects with alpha-1-anti-trypsin (AAT) deficiency by comparing AUC from Day 0 to Day 7 of plasma Alpha1-PI measured by the functional activity (potency) assay. AUC from Day 0 to Day 7 was calculated at steady state at the end of the first and second 8-week treatment periods during the 16-week double-blind, crossover phase.
Time Frame: Day 0 to Day 7
Measure: Number; unit: mg*h/mL
Groups:
- Alpha-1 MP: Sequential, blinded treatment periods of Alpha-1 MP (experimental), then crossed-over to Prolastin (active comparator), followed by open-label Alpha-1 MP
- Prolastin: Sequential, blinded treatment periods of Prolastin (active comparator), then crossed-over to Alpha-1 MP (experimental), followed by open-label Alpha-1 MP
Arm/Group | Alpha-1 MP | Prolastin
Number analyzed (Participants) | 24 | 24
mg*h/mL | 155.9 [0.97 to 1.09] | 152.4 [0.97 to 1.09]
Statistical Analysis 1: Comparison: Alpha-1 MP vs Prolastin; To compare AUC 0-7 days between the two treatments (Alpha-1 MP vs. Prolastin),natural log-transformed AUC 0-7 days values were analyzed by analysis of variance (ANOVA); Test type: Non-Inferiority or Equivalence — A total sample size of 20 subjects could demonstrate comparability of an AUC(0-7days) with 90% power up to a standard deviation of 0.288 of the difference in the log scale, expected mean treatment difference of 0 (= ratio of 1), a lower equivalence limit of -0.223 (= log 0.8), upper limit of 0.223 (= log 1.25) and a one-sided alpha of 0.05 (90% CI); Geometric least square means ratio = 1.03, 90% CI [0.97 to 1.09]

ADVERSE EVENTS:
Arm/Group | Alpha-1 MP | Prolastin
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/24
Other Adverse Events (participants affected / at risk) | 3/24 | 5/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-1 MP (N=24) | Prolastin (N=24)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-1 MP (N=24) | Prolastin (N=24)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must send a draft manuscript of the publication or abstract to the sponsor thirty days in advance of submission in order to obtain approval prior to submission of the final version for publication. This will be reviewed promptly and approval will not be withheld unreasonably. In case of a difference of opinion between the sponsor and the investigator(s), the contents of the publication will be discussed in order to find a solution which satisfies both parties.